CLINICAL TRIAL: NCT04309422
Title: Correlation Between Texture Features With CT-PET 18 FDG and Overexpression of PDL1 in Non-small-cell Lung Carcinomas During the Initial Staging.
Brief Title: Texture Features and PDL1 in CT-PET 18 FDG
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0623
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Correlation between overexpression of PDL1; texture features; CT-PET 18 FDG; Non Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overexpression of PDL1: Overexpression of PDL1
- Absence of overexpression of PDL1: Absence of overexpression of PDL1

SUMMARY:
Search correlation between texture features in CT-PET 18 FDG and overexpression of PDL1 in non-small cell lung carcinomas during the inital staging.

The hypothesis is that overexpression of PDL1is correlated with at least one texture feature among those selected.

84 CT-PET 18 FDG at the initial staging of a non small cell lung carcinoma (adenocarcinoma or squamous cell carcinoma), whose the biopsed site was the primitive site or the drainage lymphadenopathy, without previous treatment, were recruited and analyzed by a software allowing to estimate texture features.

ELIGIBILITY:
Inclusion criteria:

* adult patient ;
* first CT-PET 18 FDG realized for the inital staging ;
* absence of previous treatment for a thoracic neoplasm ;
* biopsy realized on the primitive site or local drainage lymphadenopathy ;
* primitive site viewable with morphological imagery ;
* availability of evaluation of PDL1's overexpression ;

Exclusion criteria

- Refusal to participate in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with initial CT-PET 18 FDG realized in the nuclear service of Montpellier university hospital, with non small cell lung carcinoma diagnosed with biopsy of the primitive site or local drainage lymphadenopathy.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Correlation between at least one texture feature and overexpression of PDL1 | 1 day
  Correlation between at least one texture feature and overexpression of PDL1

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste MALLET, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC